CLINICAL TRIAL: NCT06829251
Title: The Effect of Self-Administered Ear Massage on Stress, Anxiety Levels, and Sleep Quality in Parents of Children Diagnosed With Type 1 Diabetes
Brief Title: Effect of Ear Massage on Stress, Anxiety, and Sleep Quality in Parents of Children With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ebru Koç, Master of Science in Public Health Nursing student, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinU-SBE-EK-01
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Stress; Anxiety; Sleep Quality
Keywords: Ear Massage; Stress; Anxiety; Sleep Quality; Tip-1 Diabetes Mellitus; Parents
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study is designed as a single-blind, randomized, sham-controlled, interventional research to determine the effect of self-administered effective ear massage on stress, anxiety levels, and sleep quality in parents of children diagnosed with Type 1 diabetes. Participants in the intervention group will perform effective ear massage, while participants in the control group will receive sham ear massage that mimics the intervention but does not stimulate pressure points.
Who Masked: Participant
Masking Description: The parents participating in the study will not know which group they are in. During the statistical analysis of the study, group codes will be created as A and B, and which codes represent which groups will be kept in a sealed envelope by a researcher who is not involved in the analysis phase. The group codes will be revealed after all analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effective Ear Massage Group (Experimental): Parents in this group will receive a 20-minute individual instruction on ear massage via WhatsApp (What's up Application). They will be taught an effective ear massage technique targeting key stress, anxiety, and sleep points. The massage will be performed on the entire ear with varying pressure over a 3-minute period. During the sessions, parents will be assessed using the Readiness for Intervention Form . When the massage starts the day after the interview, parents will fill out the Ear Massage Follow-Up Form , and a reminder message will be sent by the researcher before the scheduled massage time, asking parents to set an alarm on their phones. Additionally, the Ear Massage Training Brochure will be provided. After two weeks, the Depression, Anxiety, Stress Scale-21 (DASS-21) and Pittsburgh Sleep Quality Index will be administered. At the end of the study, parents will be reminded to consider psychiatric clinic consultations.
  Interventions: Behavioral: Effective Ear Massage
- Sham Ear Massage Group (Sham Comparator): Parents in this group will receive 20-minute individual instruction on ear massage via WhatsApp (What's up Application). They will perform a sham ear massage on the helix outer rim,helix crest and points 1, 2, and 3 without applying pressure. This 1-minute sham massage mimics the intervention but does not affect stress, anxiety, or sleep. Parents will be assessed using the Readiness for Intervention Form. The massage will start the day after the interview. Parents will fill out the Ear Massage Follow-Up Form . A reminder will be sent by the researcher before the massage time, asking them to set an alarm. Additionally, the Ear Massage Training Brochure will be provided. After two weeks, the Depression, Anxiety, Stress Scale-21 (DASS-21) and Pittsburgh Sleep Quality Index will be administered. The sham control group will later learn the effective ear massage technique. At the end, parents will be reminded to consider psychiatric consultations.
  Interventions: Behavioral: Sham Ear Massage

INTERVENTIONS:
Behavioral: Effective Ear Massage — The intervention consists of a structured ear massage technique administered daily for 2 weeks. Parents will receive training on how to target specific pressure points on the ear to reduce stress and anxiety, and improve sleep quality. This training will be conducted via WhatsApp (What's up Application) for 20 minutes, followed by daily massage practice. The massage will be performed using varying pressure over a 3-minute period on the entire ear, focusing on stress and sleep points.
  Arms: Effective Ear Massage Group
Behavioral: Sham Ear Massage — The sham intervention involves a 1-minute ear massage on the outer helix rim, helix crest, and helix points 1, 2, and 3, without applying any pressure. The goal of the sham massage is to mimic the process of ear massage while ensuring no physiological effect on stress, anxiety, or sleep quality.
  Arms: Sham Ear Massage Group

SUMMARY:
The purpose of this clinical trial is to determine the effect of self-administered ear massage on stress, anxiety levels, and sleep quality in parents of children diagnosed with Type 1 diabetes. Additionally, it aims to assess whether ear massage can prevent stress, anxiety, and poor sleep quality. The primary questions it seeks to answer are:

H0: There is no significant difference in the mean stress scores between the intervention and control groups of parents.

H0: There is no significant difference in the mean anxiety scores between the intervention and control groups of parents.

H0: There is no significant difference in the mean Pittsburgh Sleep Quality Index (PSQI) scores between the intervention and control groups of parents.

Researchers will compare the effects of ear massage on stress, anxiety levels, and sleep quality with a sham control.

Participants:

Intervention group: Self-administered effective ear massage twice daily for two weeks, with each session lasting three minutes, totaling 28 sessions.

Control group: Self-administered sham ear massage twice daily for two weeks, with each session lasting one minute, totaling 28 sessions.

Parents will be reached by sending an invitation letter to the groups they are in on WhatsApp (What's up Application) and Instagram.Volunteer parents will be evaluated for their eligibility criteria and assessed using the 'Depression, Anxiety, Stress Scale-21 (DASS-21)' form. Suitable parents will be sent the informed consent form, personal information form, and 'Pittsburgh Sleep Quality Index'. After the initial data collection, an online ear massage training will be provided. Both groups will receive a 20-minute individual online ear massage training. The Readiness Assessment Form will be used during the training. The application will start the next day. During the implementation process, brochures and video support will be provided by the researcher, and reminder messages will be sent at the times of application. Additionally, participants will be asked to set reminder alarms on their phones. Participants will complete the Ear Massage Tracking Form during the implementation process. At the end of the two-week period, the 'Depression, Anxiety, Stress Scale-21 (DASS-21)' form and the 'Pittsburgh Sleep Quality Index' will be filled out.

DETAILED DESCRIPTION:
Type 1 diabetes is a chronic metabolic disease characterized by insulinopenia and hyperglycemia, resulting from the destruction of pancreatic beta cells responsible for insulin production due to autoimmune or non-autoimmune causes in the childhood group [1]. Since Type 1 diabetes is mostly diagnosed at a young age, parents have significant responsibilities in the management and care of Type 1 diabetes [2]. The need for continuous 24-hour care leads to parents being detached from their social life, experiencing increased stress and anxiety levels, and reduced sleep quality [2]. Research indicates that approximately 20% to 30% of parents of children diagnosed with Type 1 diabetes report clinically significant stress (life stress or parenting stress), anxiety, depression, and post-traumatic stress symptoms [3,4, 5]. Additionally, studies have shown that 76% of parents experience clinically significant sleep disorders [6].

When parents cannot cope adequately with increased stress, they experience physiological, psychological, behavioral, social, and cognitive problems [7]. Non-pharmacological methods used to cope with stress include cognitive-behavioral therapies, yoga, breathing exercises, massage, acupressure, and acupuncture. Another method that meets the criteria of accessibility, reliability, cost-effectiveness, and self-applicability among non-pharmacological methods used to cope with experienced stress is ear massage [8]. According to Traditional Chinese Medicine, the ear is directly or indirectly connected to twelve meridians, and stimulating the ear restores balance between vital energy (qi) and blood flow yin-yang [9]. There are reflex points on these meridians that stimulate internal organs and qi to relieve stress, anxiety, and reduce sleep problems [10]. These reflex points are points on the body's surface through which the qi of internal organs and meridians pass. Each point is associated with specific psychological, neurological, and immunological effects to best balance physiological and psychological functions [11].

Furthermore, the only peripheral branch of the vagus nerve is in the outer ear. Stimulation of the auricular vagus nerve suppresses the sympathetic nerve and activates the parasympathetic nerve [12]. Decreased sympathetic and increased parasympathetic activity helps reduce stress levels and stress-related anxiety by lowering cortisol and epinephrine levels [13]. Decreased cortisol levels increase melatonin levels, promoting sleep and relaxation [14]. Compared to acupuncture and ear acupressure, ear massage has the advantage of being tool-free and easy to apply. It can also be easily applied by individuals with temporal, spatial, and situational constraints. Since it does not involve any invasive intervention, it has no side effects [8].

Due to these features, it has the potential to be widely used by nurses to reduce patients' stress, anxiety, and sleep problems in clinical and field settings, and according to nursing regulations, massage is one of the independent roles of nurses [15, 16]. Complementary and alternative treatments involving ear massage are observed to have fewer clinical studies and a lack of scientific evidence compared to modern medicine; therefore, a validation process through scientific research experiments is needed [12].

Ear massage is a promising, easily applicable, non-invasive, safe, and cost-effective non-pharmacological method for reducing stress and anxiety symptoms experienced by caregiver family members and increasing sleep quality. However, more evidence is needed regarding the effectiveness of ear massage [8, 12]. This study aims to determine the effect of ear massage on stress, anxiety levels, and sleep quality in parents of children diagnosed with Type 1 diabetes [8].

ELIGIBILITY:
Inclusion Criteria:

Between February 2025 and July 2025, parents of children diagnosed with Type 1 diabetes, who are registered in the Mersin Diabetics group on WhatsApp (What's up Application), the Type 1 Diabetics association on Instagram, and the community forums and groups of diabetes education nurses and dietitians, will be eligible to participate in the study.

* Those who are willing to participate in the study and have signed the informed consent form
* Those who score medium or higher [stress (10 points or more) or anxiety (8 points or more)] on the Depression, Anxiety, Stress Scale-21 (DASS-21) and prefer to perform ear massage first over immediately receiving psychiatric support
* Those who have the facilities to participate in online training (internet, phone/tablet/computer, etc.) will be included in the sample.

Exclusion Criteria:

Between February 2025 and July 2025, parents of children diagnosed with Type 1 diabetes, who are registered in the Mersin Diabetics group on WhatsApp (What's up Application), the Type 1 Diabetics association on Instagram, and the community forums and groups of diabetes education nurses and dietitians, will be eligible to participate in the study.

* Those who are not willing to participate in the study
* Those with a psychiatric diagnosis made by a doctor
* Those who score medium or higher [stress (10 points or more) or anxiety (8 points or more)] on the DASS-21 scale, but prefer to receive psychiatric support first over ear massage after immediately receiving psychiatric support
* Those receiving regular professional psychological support
* Those taking antidepressants, anticonvulsants, or sleeping pills
* Pregnant women or those suspected of being pregnant
* Those with auricular aplasia or hypoplasia
* Those with active infection or disruption of skin integrity in the ear area (ulcer, eczema, urticaria, surgical incision, etc.)
* Those with visual, hearing, or speech impairments
* Those receiving regular complementary or alternative treatments for stress, anxiety, and sleep (acupuncture, facial massage, phytotherapy, meditation, breathing exercises, etc.) will not be included in the sample.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Stress Levels | 2 weeks (after intervention)
  Changes in stress levels will be measured at two weeks using the Depression, Anxiety, Stress Scale-21 (DASS-21). Lovibond (1995) developed the original 42-item scale, and the same authors later created the 21-item short form, which was adapted to Turkish culture by Sarıçam (2018). The scale consists of seven items each for evaluating depression, anxiety, and stress. Responses are given on a 4-point Likert scale (0 = Never, 3 = Always). The Cronbach's Alpha coefficients of the scale are 0.87 for depression, 0.85 for anxiety, and 0.81 for stress.
  Depression is classified as follows: (0-4) Normal, (5-6) Mild, (7-10) Moderate, (11-13) Severe, (14+) Extremely Severe Depression. Anxiety is classified as: (0-3) Normal, (4-5) Mild, (6-7) Moderate, (8-9) Severe, (10+) Extremely Severe Anxiety. Stress is classified as: (0-7) Normal, (8-9) Mild, (10-12) Moderate, (13-16) Severe, (17+) Extremely Severe Stress.Only the stress and anxiety subscales will be assessed.
Change in Anxiety Levels | 2 weeks (after intervention)
  Changes in anxiety levels will be measured at two weeks using the Depression, Anxiety, Stress Scale-21 (DASS-21). Lovibond (1995) developed the original 42-item scale, and the same authors later created the 21-item short form, which was adapted to Turkish culture by Sarıçam (2018). The scale consists of seven items each for evaluating depression, anxiety, and stress. Responses are given on a 4-point Likert scale (0 = Never, 3 = Always). The Cronbach's Alpha coefficients of the scale are 0.87 for depression, 0.85 for anxiety, and 0.81 for stress. Depression is classified as follows: (0-4) Normal, (5-6) Mild, (7-10) Moderate, (11-13) Severe, (14+) Extremely Severe Depression. Anxiety is classified as: (0-3) Normal, (4-5) Mild, (6-7) Moderate, (8-9) Severe, (10+) Extremely Severe Anxiety. Stress is classified as: (0-7) Normal, (8-9) Mild, (10-12) Moderate, (13-16) Severe, (17+) Extremely Severe Stress.Only the stress and anxiety subscales will be assessed.
Change in Sleep Quality | 2 weeks (after intervention)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 24-item questionnaire. The Pittsburgh Sleep Quality Index was developed by Buysse et al. in 1989 to assess sleep quality in psychiatric practice and clinical research. The PSQI evaluates sleep quality over the past month. The validity and reliability studies of this scale for the Turkish culture were conducted by Ağargün et al. in 1996, and the Cronbach's alpha reliability coefficient of the scale was found to be 0.80.Nineteen questions are self-reported, and the last 5 questions are answered by a spouse or roommate. Eighteen items are included in the scoring and are grouped into 7 component scores. Each item is rated on a scale of 0-3. The total score ranges from 0-21, with higher scores indicating poorer sleep quality.

SECONDARY OUTCOMES:
Change in Energy Levels | Every day (for 2 weeks).
  Participants' daily energy levels will be assessed using a rating scale of '0 Very Low' to '10 Very High'. Changes in energy levels will be tracked daily and recorded in the massage tracking form to determine the impact of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Health Sciences Institute Nursing Department Çiftlikköy Campus Yenişehir / MERSİN TURKEY, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Zhang J, Jin Y, Zhang Q. Auricular Acupressure Therapy for Patients with Cancer with Sleep Disturbance: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2021 Oct 14;2021:3996101. doi: 10.1155/2021/3996101. eCollection 2021. PMID 34691214
- [Background] Chen SR, Hou WH, Lai JN, Kwong JSW, Lin PC. Effects of Acupressure on Anxiety: A Systematic Review and Meta-Analysis. J Integr Complement Med. 2022 Jan;28(1):25-35. doi: 10.1089/jicm.2020.0256. PMID 35085025
- [Background] Park S, Park H, Bang YY. The Effects of Auricular Acupressure on Physiological Index, Depression, Anxiety, and Stress for Elders With Hypertension. Holist Nurs Pract. 2023 Jan-Feb 01;37(1):24-33. doi: 10.1097/HNP.0000000000000558. PMID 36378089
- [Background] Tseng YT, Chen IH, Lee PH, Lin PC. Effects of auricular acupressure on depression and anxiety in older adult residents of long-term care institutions: A randomized clinical trial. Geriatr Nurs. 2021 Jan-Feb;42(1):205-212. doi: 10.1016/j.gerinurse.2020.08.003. Epub 2020 Sep 11. PMID 32921508
- [Background] Cha NH, Park YK, Sok SR. Effects of Auricular Acupressure Therapy on Stress and Sleep Disturbance of Middle-Aged Women in South Korea. Holist Nurs Pract. 2017 Mar/Apr;31(2):102-109. doi: 10.1097/HNP.0000000000000197. PMID 28181975
- [Background] Kuo SY, Tsai SH, Chen SL, Tzeng YL. Auricular acupressure relieves anxiety and fatigue, and reduces cortisol levels in post-caesarean section women: A single-blind, randomised controlled study. Int J Nurs Stud. 2016 Jan;53:17-26. doi: 10.1016/j.ijnurstu.2015.10.006. Epub 2015 Oct 22. PMID 26525188
- [Background] Xin D, Cui L, Wang L, Zhang Q, Chen X, Shi Y, Zhu W, Xu N, Li W, Wang Y. Effect of auricular acupressure on sleep quality in breast cancer patients: A systematic review and meta-analysis of randomized controlled trials. Complement Ther Clin Pract. 2024 Nov;57:101876. doi: 10.1016/j.ctcp.2024.101876. Epub 2024 Jun 9. PMID 38925078
- [Background] Rechenberg K, Grey M, Sadler L. Stress and Posttraumatic Stress in Mothers of Children With Type 1 Diabetes. J Fam Nurs. 2017 May;23(2):201-225. doi: 10.1177/1074840716687543. Epub 2017 Jan 10. PMID 28795899
- [Background] Morrow T, Bhatia SH, Parmar AM, Baker L, Abadula F, Williamson D, Choudhary A, Jaser SS. Sleep Habits of Early School-Aged Children with Type 1 Diabetes and Their Parents: Family Characteristics and Diabetes Management. Behav Sleep Med. 2022 Sep-Oct;20(5):649-658. doi: 10.1080/15402002.2021.1977305. Epub 2021 Sep 24. PMID 34559603
- [Background] Bassi G, Mancinelli E, Di Riso D, Salcuni S. Parental Stress, Anxiety and Depression Symptoms Associated with Self-Efficacy in Paediatric Type 1 Diabetes: A Literature Review. Int J Environ Res Public Health. 2020 Dec 28;18(1):152. doi: 10.3390/ijerph18010152. PMID 33379307
- [Background] Horsch A, McManus F, Kennedy P, Edge J. Anxiety, depressive, and posttraumatic stress symptoms in mothers of children with type 1 diabetes. J Trauma Stress. 2007 Oct;20(5):881-91. doi: 10.1002/jts.20247. PMID 17955536
- [Background] Whittemore R, Jaser S, Chao A, Jang M, Grey M. Psychological experience of parents of children with type 1 diabetes: a systematic mixed-studies review. Diabetes Educ. 2012 Jul-Aug;38(4):562-79. doi: 10.1177/0145721712445216. Epub 2012 May 11. PMID 22581804
- [Background] Azimi T, Johnson J, Campbell SM, Montesanti S. Caregiver burden among parents of children with type 1 diabetes: A qualitative scoping review. Heliyon. 2024 Mar 12;10(6):e27539. doi: 10.1016/j.heliyon.2024.e27539. eCollection 2024 Mar 30. PMID 38524615
- See also: A comprehensive study explaining the pathophysiology, diagnosis, and management of type-1 diabetes. — https://dergipark.org.tr/tr/download/article-file/909246
- See also: Link to the Official Gazette Containing Regulations in the Regulation of the Ministry of Health of the Republic of Turkey — https://www.resmigazete.gov.tr/eskiler/2011/04/20110419-5.htm